CLINICAL TRIAL: NCT00540488
Title: Randomized, Double Blind, Three Way Crossover Comparison of Glucose and Insulin Responses During a Meal Glucose Tolerance Test in Subjects With Type 2 Diabetes Consuming Disease-Specific Versus Standard Nutritional Formula
Brief Title: Glucose/Insulin Responses:Subjects With Type 2 Diabetes Consuming Diabetes-Specific vs Standard Nutritional Formulas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRDB09
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2007-10-15 (Estimated); Status verified 2007-10

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Other: Adult enteral formula

SUMMARY:
To measure and compare the glycemic and insulinemic responses of subjects consuming a standard and two diabetes-specific products.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent
* 18-75 years of age
* history of type 2 diabetes
* males and non-pregnant, non-lactating females

Exclusion Criteria:

* subject uses insulin for glucose control
* significant cardiovascular event <12 weeks prior to study entry
* active malignancies
* history of end stage renal disease
* history of organ transplant
* current hepatic disease
* intervention for HIB
* takes niacin
* history of gastroparesis
* active disease that may interfere with nutrient intake
* allergy or intolerance to ingredients in the study products

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2002-08

PRIMARY OUTCOMES:
Adjusted area under the curve (adj-AUC) of glucose response | 0-240 minutes

SECONDARY OUTCOMES:
Adjusted peak for glucose and insulin response;peak time for glucose and insulin response; Adj-AUC for insulin response; change in glucose and insulin; subjective gastrointestinal tolerance | 0 - 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Alish, PhD, Study Chair — Abbott Nutrition
Locations (2):
- United States (2):
  - Protocare Trials, Chicago Center for Clinical Research, Chicago, Illinois
  - Medical University of South Carolina, Charleston, North Carolina